CLINICAL TRIAL: NCT00188461
Title: Dose Reduction in Thoracic CT: A Comparison of on Line Automatic Dose Reduction and a 50% Reduction in Dose
Brief Title: Dose Reduction in Thoracic CT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 03-0875
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2007-04-23 (Estimated); Status verified 2005-09

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

INTERVENTIONS:
Device: CT Thorax

SUMMARY:
Hypothesis: Does a 50% reduction in radiation in dose significantly affect the diagnostic quality of chest CT

DETAILED DESCRIPTION:
Patients with Lymphoma are recruited and have a follow up CT performed at 50% of the standard exposure parameters. The studies are compared for image quality with a recent (<3 months) thoracic CT performed at standard exposure parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Lymphoma

Exclusion Criteria:

* No recent (<3 months) thoracic CT

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2004-01; Study Completion 2005-08

PRIMARY OUTCOMES:
Evaluating the diagnostic quality of thoracic CT exams performed at 50% of standard dose parameters

CONTACTS AND LOCATIONS:
Overall Officials: Narinder Paul, FRCP C, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada